CLINICAL TRIAL: NCT05064449
Title: A Phase 1, Open-Label Study to Evaluate the Effect of Itraconazole and Mefenamic Acid on the Single-Dose Pharmacokinetic Profile of Soticlestat in Healthy Participants
Brief Title: A Study of Soticlestat With Itraconazole and Mefenamic Acid in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: TAK-935-1007
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Results first posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2022-11

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy
MeSH Terms: interventions — soticlestat; Itraconazole; Mefenamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part 1: Soticlestat 300 mg + Itraconazole 200 mg (Experimental): Soticlestat 300 milligram (mg), tablets, orally, once on Day 1 in Period 1, followed by 4 days washout period, followed by itraconazole 200 mg solution, orally, once daily from Day 1 up to Day 11, further followed by soticlestat 300 mg tablet, orally along with itraconazole 200 mg solution, orally on the morning of Day in Period 2.
  Interventions: Drug: Soticlestat; Drug: Itraconazole
- Part 2: Soticlestat 300 mg + Mefenamic Acid 500 mg (Experimental): Soticlestat 300 mg, tablets, orally, once on Day 1 in Period 1, followed by 4 days washout period, followed by single dose of mefenamic acid 500 mg capsule (first dose only), orally on the morning of Day 1 and 250 mg subsequent doses at every six hours up to Day 7 in Period 2, further followed by soticlestat 300 mg tablet, orally, followed by mefenamic acid 250 mg capsule, orally in morning of Day 2 in Period 2.
  Interventions: Drug: Soticlestat; Drug: Mefenamic acid

INTERVENTIONS:
Drug: Soticlestat — Soticlestat tablets.
  Other Names: TAK-935
Drug: Itraconazole — Itraconazole oral solution.
  Arms: Part 1: Soticlestat 300 mg + Itraconazole 200 mg
Drug: Mefenamic acid — Mefenamic acid capsule.
  Arms: Part 2: Soticlestat 300 mg + Mefenamic Acid 500 mg

SUMMARY:
The main aim of this study is to check how itraconazole and mefenamic acid affect the way soticlestat is processed by the body.

The study will have 2 parts. Participants can only participate in one study part.

Part 1: Participants will check into the study clinic to receive soticlestat, four days later they will begin receiving itraconazole and will stay in the clinic for 11 more days, receiving soticlestat in combination with itraconazole on one of those days. Participants will be contacted about 8 days after leaving the clinic for follow-up.

Part 2: Participants will check into the study clinic to receive soticlestat, four days later they will begin receiving mefenamic acid and will stay in the clinic for 7 more days, receiving soticlestat in combination with mefenamic acid on one of those days.. Participants will be contacted about 9 days after leaving the clinic for follow-up.

DETAILED DESCRIPTION:
The drug being tested in this study is called soticlestat (TAK-935). The study will evaluate the safety and tolerability of soticlestat when co-administered with either itraconazole or mefenamic acid in healthy participants.

The study will be conducted in 2 parts: Part 1 (drug-drug interaction [DDI] with itraconazole), Part 2 (DDI with mefenamic acid). The study will enroll approximately 28 participants. Participants will be enrolled into two parts (Part 1 and Part 2) to receive soticlestat along with adjunctive therapy itraconazole and mefenamic acid as:

* Part 1: Soticlestat 300 mg + Itraconazole 200 mg
* Part 2: Soticlestat 300 mg + Mefenamic Acid 500 mg (first dose only) and 250 mg (subsequent doses)

Both Parts 1 and 2 will have two period (Periods 1 and 2). In Period 1, participants will receive only soticlestat (study drug) and in Period 2, participants will receive study drug along with either itraconazole or mefenamic acid depending upon in which part they are in. The data will be collected and stored in electronic case report form (eCRF).

This single-center trial will be conducted in the United States. The overall duration of the study is approximately 52 days for participants in Part 1 (includes screening and follow-up), but 48 days for participants in Part 2 (including screening and follow-up). There will be follow up for all participants approximately 15 days after the last dose of soticlestat in each study part.

ELIGIBILITY:
Inclusion Criteria:

1. Has body mass index (BMI) greater than or equal to (>=) 18.0 and less than or equal to (<=) 32.0 kilogram per meter square (kg/m^2) at screening.
2. Continuous non-smoker who has not used nicotine-containing products for at least 90 days prior to the first dosing.
3. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or electrocardiograms (ECGs), as deemed by the Investigator or designee.

   * Supine blood pressure is >=90/40 millimeter of mercury (mmHg) and <=140/90 mmHg at screening;
   * Supine pulse rate is >=45 beats per minute (bpm) and <=100 bpm at screening;
   * QT interval corrected for pulse rate using Fridericia's formula (QTcF) is <=450 millisecond (msec) (males) or <=470 msec (females) and ECG findings considered normal or not clinically significant by the Investigator or designee at screening;
   * Estimated creatinine clearance >=80 milliliter per minute (mL/min) at screening;
   * Liver function tests including alanine aminotransferase (ALT) or aspartate aminotransferase (AST) <=1.5*the upper limit of normal (ULN) at screening and check-in.
4. Able to swallow multiple tablets.

Exclusion Criteria:

1. Has history of any illness that, in the opinion of the Investigator or designee, might confound the results of the study or poses an additional risk to the participants by their participation in the study.
2. Has history or presence of alcoholism or drug abuse within the past 2 years prior to the first dosing.
3. Has history or presence of hypersensitivity or idiosyncratic reaction to the study drugs or related compounds.
4. Unable to refrain from or anticipates the use of:

   • Any drug, including prescription and non-prescription medications, herbal remedies, or vitamin supplements within 14 days prior to the first dosing. Thyroid hormone replacement medication may be permitted if the participant has been on the same stable dose for the immediate 3 months prior to first dosing.
5. Has history of alcohol consumption exceeding 2 standard drinks per day on average (1 glass is approximately equivalent to the following: beer 354 milliliter (mL)/12 Ounce [oz], wine [118 mL/4 oz], or distilled spirits [29.5 mL/1 oz] per day).
6. Consumes excessive amounts, defined as greater than 4 servings (1 serving is approximately equivalent to 120 mg of caffeine), of coffee, tea, cola, energy drinks, or other caffeinated beverages per day.
7. Has been on a diet incompatible with the on-study diet, in the opinion of the Investigator or designee, within the 30 days prior to the first dosing and throughout the study.
8. Donation of blood or significant blood loss within 56 days prior to the first dosing.
9. Plasma donation within 7 days prior to the first dosing.
10. Has participation in another clinical study within 30 days or 5 half-lives prior to the first dosing. The 30-day window or 5 half-lives will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of Period 1 of the current study.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2021-11-21 (Actual); Study Completion 2021-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/6165afd6eb0e19002afd68c4

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 14 October 2021 to 30 November 2021.
Pre-assignment Details: Healthy participants were enrolled in this 2-part study to receive soticlestat tablets alone in Period 1 and soticlestat tablets and itraconazole solution in Period 2 of Part 1; and soticlestat tablets alone in Period 1 and soticlestat tablets and mefenamic acid capsules in Period 2 of Part 2. Both study parts (Parts 1 and 2) were conducted independently from one another, no crossover happened between both parts.
Groups:
- Part 1: Soticlestat 300 mg + Itraconazole 200 mg: Soticlestat 300 milligram (mg) administered as 3*100 mg tablets, orally, once on Day 1 of Period 1, followed by 4 days washout period, further followed by itraconazole 200 mg administered as 20 milliliter (mL) of 10 milligram per milliliter (mg/ml) solution, orally, once daily from Day 1 up to Day 11 of Period 2 and soticlestat 300 mg administered as 3*100 mg tablets, orally, once on Day 5 of Period 2.
- Part 2: Soticlestat 300 mg + Mefenamic Acid 500 mg and 250 mg: Soticlestat 300 mg administered as 3*100 mg tablets, orally, once on Day 1 of Period 1, followed by 4 days washout period, further followed by initial single dose of mefenamic acid 500 mg administered as 2*250 mg capsules, orally on the morning of Day 1 and 250 mg subsequent doses at every six hours from Day 1 up to Day 7 of Period 2, and soticlestat 300 mg administered as 3*100 mg tablets, orally, once on Day 2 of Period 2.
Period: Period 1 (1 Day)
Arm/Group | Part 1: Soticlestat 300 mg + Itraconazole 200 mg | Part 2: Soticlestat 300 mg + Mefenamic Acid 500 mg and 250 mg
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0
Period: Washout Period (4 Days)
Arm/Group | Part 1: Soticlestat 300 mg + Itraconazole 200 mg | Part 2: Soticlestat 300 mg + Mefenamic Acid 500 mg and 250 mg
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0
Period: Period 2(Part 1:Day 1-12;Part 2:Day 1-8)
Arm/Group | Part 1: Soticlestat 300 mg + Itraconazole 200 mg | Part 2: Soticlestat 300 mg + Mefenamic Acid 500 mg and 250 mg
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of the study drug(s) were included in the safety analysis set.
Groups:
- Part 1: Soticlestat 300 mg + Itraconazole 200 mg: Soticlestat 300 mg administered as 3*100 mg tablets, orally, once on Day 1 of Period 1, followed by 4 days washout period, further followed by itraconazole 200 mg administered as 20 mL of 10 mg/ml solution, orally, once daily from Day 1 up to Day 11 of Period 2 and soticlestat 300 mg administered as 3*100 mg tablets, orally, once on Day 5 of Period 2.
- Total: Total of all reporting groups
Arm/Group | Part 1: Soticlestat 300 mg + Itraconazole 200 mg | Part 2: Soticlestat 300 mg + Mefenamic Acid 500 mg and 250 mg | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 28
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 11 | 12 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 2
  Black or African American | 4 | 5 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White | 8 | 5 | 13
  White, American Indian or Alaska Native | 0 | 1 | 1
  White, Black or African American | 0 | 1 | 1
  White, Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States of America | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Part 1, Cmax: Maximum Observed Plasma Concentration for Soticlestat When Administered Alone and With Itraconazole
Time Frame: Soticlestat alone: Period 1, Day 1 pre-dose and at multiple timepoints (up to 96 hours) post-dose; Soticlestat with itraconazole: Period 2, Day 5 pre-dose and at multiple timepoints (up to 168 hours) post-dose
Population: All participants who complied sufficiently with the protocol and display an evaluable pharmacokinetic (PK) profile (example, exposure to treatment, availability of measurements and absence of major protocol violations) were included in the PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Part 1: Soticlestat 300 mg Alone: Soticlestat 300 mg administered as 3*100 mg tablets, orally, once on Day 1 of Period 1.
- Part 1: Soticlestat 300 mg + Itraconazole 200 mg: Itraconazole 200 mg administered as 20 mL of 10 mg/ml solution, orally, once daily from Day 1 up to Day 11 of Period 2, and soticlestat 300 mg administered as 3*100 mg tablets, orally, once on Day 5 of Period 2.
Arm/Group | Part 1: Soticlestat 300 mg Alone | Part 1: Soticlestat 300 mg + Itraconazole 200 mg
Number analyzed (Participants) | 14 | 14
nanogram per milliliter (ng/mL) | 1310 (80.2) | 1527 (65.5)
Statistical Analysis 1: Comparison: Part 1: Soticlestat 300 mg Alone vs Part 1: Soticlestat 300 mg + Itraconazole 200 mg; Linear mixed-effects model was used for analysis, using fixed-effect (treatment), random-effect (participants). The point estimates and the 90 percent (%) confidence intervals (CIs) for the geometric mean ratio (GMR) of Cmax for soticlestat with versus without itraconazole were calculated by exponentiation of the point estimates of the differences between treatments and the corresponding 90% CIs from the analyses on the ln-transformed Cmax; Test type: Other; Geometric Mean Ratio (%) = 116.59, 90% CI 2-sided [91.30 to 148.90] — GMR (%) was calculated as 100*(Soticlestat + Itraconazole / Soticlestat Alone)

2. Primary Outcome: Part 2, Cmax: Maximum Observed Plasma Concentration for Soticlestat When Administered Alone and With Mefenamic Acid
Time Frame: Soticlestat alone: Period 1, Day 1 pre-dose and at multiple timepoints (up to 96 hours) post-dose; Soticlestat with mefenamic acid: Period 2, Day 2 pre-dose and at multiple timepoints (up to 144 hours) post-dose
Population: All participants who complied sufficiently with the protocol and display an evaluable PK profile (example, exposure to treatment, availability of measurements and absence of major protocol violations) were included in the PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part 2: Soticlestat 300 mg Alone: Soticlestat 300 mg administered as 3*100 mg tablets, orally, once on Day 1 of Period 1.
- Part 2: Soticlestat 300 mg + Mefenamic Acid 500 mg and 250 mg: Initial single dose of mefenamic acid 500 mg administered as 2*250 mg capsules, orally on the morning of Day 1 and 250 mg subsequent doses at every six hours from Day 1 up to Day 7, and soticlestat 300 mg administered as 3*100 mg tablets, orally, once on Day 2 of Period 2.
Arm/Group | Part 2: Soticlestat 300 mg Alone | Part 2: Soticlestat 300 mg + Mefenamic Acid 500 mg and 250 mg
Number analyzed (Participants) | 14 | 14
ng/mL | 1414 (58.4) | 1517 (55.8)
Statistical Analysis 1: Comparison: Part 2: Soticlestat 300 mg Alone vs Part 2: Soticlestat 300 mg + Mefenamic Acid 500 mg and 250 mg; Linear mixed-effects model was used for analysis, using fixed-effect (treatment), random-effect (participants). The point estimates and the 90% CIs for the GMR of Cmax for soticlestat with versus without mefenamic acid were calculated by exponentiation of the point estimates of the differences between treatments and the corresponding 90% CIs from the analyses on the ln-transformed Cmax; Test type: Other; Geometric Mean Ratio (%) = 107.31, 90% CI 2-sided [88.02 to 130.83] — GMR (%) was calculated as 100*(Soticlestat + Mefenamic Acid / Soticlestat Alone)

3. Primary Outcome: Part 1, AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Soticlestat When Administered Alone and With Itraconazole
Time Frame: as for outcome 1
Population: All participants who complied sufficiently with the protocol and display an evaluable PK profile (example, exposure to treatment, availability of measurements and absence of major protocol violations) were included in the PK analysis set. Here, "overall number of participants analyzed" signified those who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hours per milliliter(ng*hr/mL)
Arm/Group | Part 1: Soticlestat 300 mg Alone | Part 1: Soticlestat 300 mg + Itraconazole 200 mg
Number analyzed (Participants) | 12 | 9
nanogram*hours per milliliter(ng*hr/mL) | 1483 (56.1) | 1914 (42.8)
Statistical Analysis 1: Comparison: Part 1: Soticlestat 300 mg Alone vs Part 1: Soticlestat 300 mg + Itraconazole 200 mg; Linear mixed-effects model was used for analysis, using fixed-effect (treatment), random-effect (participants). The point estimates and the 90% CIs for the GMR of AUC∞ for soticlestat with versus without itraconazole were calculated by exponentiation of the point estimates of the differences between treatments and the corresponding 90% CIs from the analyses on the ln-transformed AUC∞; Test type: Other; Geometric Mean Ratio (%) = 123.96, 90% CI 2-sided [106.21 to 144.68] — GMR (%) was calculated as 100*(Soticlestat + Itraconazole / Soticlestat Alone)

4. Primary Outcome: Part 2, AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Soticlestat When Administered Alone and With Mefenamic Acid
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 2: Soticlestat 300 mg Alone | Part 2: Soticlestat 300 mg + Mefenamic Acid 500 mg and 250 mg
Number analyzed (Participants) | 11 | 9
ng*hr/mL | 1533 (42.2) | 1594 (45.6)
Statistical Analysis 1: Comparison: Part 2: Soticlestat 300 mg Alone vs Part 2: Soticlestat 300 mg + Mefenamic Acid 500 mg and 250 mg; Linear mixed-effects model was used for analysis, using fixed-effect (treatment), random-effect (participants). The point estimates and the 90% CIs for the GMR of AUC∞ for soticlestat with versus without mefenamic acid were calculated by exponentiation of the point estimates of the differences between treatments and the corresponding 90% CIs from the analyses on the ln-transformed AUC∞; Test type: Other; Geometric Mean Ratio (%) = 100.57, 90% CI 2-sided [86.17 to 117.38] — GMR (%) was calculated as 100*(Soticlestat + Mefenamic Acid / Soticlestat Alone)

5. Primary Outcome: Part 1, AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Soticlestat When Administered Alone and With Itraconazole
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 1: Soticlestat 300 mg Alone | Part 1: Soticlestat 300 mg + Itraconazole 200 mg
Number analyzed (Participants) | 14 | 14
ng*hr/mL | 1391 (54.9) | 1697 (45.3)
Statistical Analysis 1: Comparison: Part 1: Soticlestat 300 mg Alone vs Part 1: Soticlestat 300 mg + Itraconazole 200 mg; Linear mixed-effects model was used for analysis, using fixed-effect (treatment), random-effect (participants). The point estimates and the 90% CIs for the GMR of AUClast for soticlestat with versus without itraconazole were calculated by exponentiation of the point estimates of the differences between treatments and the corresponding 90% CIs from the analyses on the ln-transformed AUClast; Test type: Other; Geometric Mean Ratio (%) = 121.97, 90% CI 2-sided [103.47 to 143.79] — GMR (%) was calculated as 100*(Soticlestat + Itraconazole / Soticlestat Alone)

6. Primary Outcome: Part 2, AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Soticlestat When Administered Alone and With Mefenamic Acid
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 2: Soticlestat 300 mg Alone | Part 2: Soticlestat 300 mg + Mefenamic Acid 500 mg and 250 mg
Number analyzed (Participants) | 14 | 14
ng*hr/mL | 1423 (41.6) | 1528 (46.2)
Statistical Analysis 1: Comparison: Part 2: Soticlestat 300 mg Alone vs Part 2: Soticlestat 300 mg + Mefenamic Acid 500 mg and 250 mg; Linear mixed-effects model was used for analysis, using fixed-effect (treatment), random-effect (participants). The point estimates and the 90% CIs for the GMR of AUClast for soticlestat with versus without mefenamic acid were calculated by exponentiation of the point estimates of the differences between treatments and the corresponding 90% CIs from the analyses on the ln-transformed AUClast; Test type: Other; Geometric Mean Ratio (%) = 107.38, 90% CI 2-sided [91.68 to 125.77] — GMR (%) was calculated as 100*(Soticlestat + Mefenamic Acid / Soticlestat Alone)

7. Primary Outcome: Part 1, Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Soticlestat When Administered Alone and With Itraconazole
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | Part 1: Soticlestat 300 mg Alone | Part 1: Soticlestat 300 mg + Itraconazole 200 mg
Number analyzed (Participants) | 14 | 14
hour | 0.500 [0.50 to 0.76] | 0.503 [0.50 to 1.00]
Statistical Analysis 1: Comparison: Part 1: Soticlestat 300 mg Alone vs Part 1: Soticlestat 300 mg + Itraconazole 200 mg; Test type: Other; p = 0.2305, Wilcoxon Signed Rank Test; Median Difference (Final Values) = 0.003, 90% CI 2-sided [-0.001 to 0.126] — Difference was calculated as (Soticlestat + Itraconazole) - Soticlestat Alone. The difference of medians (treatment effect) and the corresponding 90% CI was estimated using the Hodges-Lehmann method and Walsh Averages

8. Primary Outcome: Part 2, Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Soticlestat When Administered Alone and With Mefenamic Acid
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | Part 2: Soticlestat 300 mg Alone | Part 2: Soticlestat 300 mg + Mefenamic Acid 500 mg and 250 mg
Number analyzed (Participants) | 14 | 14
hour | 0.505 [0.50 to 1.50] | 0.522 [0.51 to 0.56]
Statistical Analysis 1: Comparison: Part 2: Soticlestat 300 mg Alone vs Part 2: Soticlestat 300 mg + Mefenamic Acid 500 mg and 250 mg; Test type: Other; p = 0.5830, Wilcoxon Signed Rank Test; Median Difference (Final Values) = -0.096, 90% CI 2-sided [-0.128 to 0.018] — Difference was calculated as (Soticlestat + Mefenamic Acid) - Soticlestat Alone. The difference of medians (treatment effect) and the corresponding 90% was estimated using the Hodges-Lehmann method and Walsh Averages

9. Secondary Outcome: Parts 1 and 2: Number of Participants Reported One or More Treatment-emergent Adverse Event (TEAE)
Time Frame: Part 1: from Day 1 of Period 1 up to 15 days after the last dose of soticlestat in Period 2 (up to Day 20 in Period 2); Part 2: from Day 1 of Period 1 up to 15 days after the last dose of soticlestat in Period 2 (up to Day 17 in Period 2)
Population: All participants who received at least one dose of the study drug(s) were included in the safety analysis set.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Itraconazole 200 mg Alone: Itraconazole 200 mg administered as 20 mL of 10 mg/ml solution, orally, once daily from Day 1 up to Day 11 of Period 2.
- Part 2: Mefenamic Acid 500 mg and 250 mg: Initial single dose of mefenamic acid 500 mg administered as 2*250 mg capsules, orally on the morning of Day 1 and 250 mg subsequent doses at every six hours from Day 1 up to Day 7 of Period 2.
Arm/Group | Part 1: Soticlestat 300 mg Alone | Part 1: Itraconazole 200 mg Alone | Part 1: Soticlestat 300 mg + Itraconazole 200 mg | Part 2: Soticlestat 300 mg Alone | Part 2: Mefenamic Acid 500 mg and 250 mg | Part 2: Soticlestat 300 mg + Mefenamic Acid 500 mg and 250 mg
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14
Participants | 1 | 2 | 3 | 1 | 0 | 3

10. Secondary Outcome: Parts 1 and 2: Number of Participants With Clinically Significant Abnormal Values for Laboratory Evaluations
Time Frame: Part 1: Day 1 of Period 1 up to Day 12 of Period 2; Part 2: Day 1 of Period 1 up to Day 8 of Period 2
Population: All participants who received at least one dose of the study drug(s) were included in the safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Soticlestat 300 mg Alone | Part 1: Itraconazole 200 mg Alone | Part 1: Soticlestat 300 mg + Itraconazole 200 mg | Part 2: Soticlestat 300 mg Alone | Part 2: Mefenamic Acid 500 mg and 250 mg | Part 2: Soticlestat 300 mg + Mefenamic Acid 500 mg and 250 mg
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14
Participants | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Parts 1 and 2: Number of Participants With Clinically Significant Abnormal Values for Vital Signs
Time Frame: Part 1: Day 1 of Period 1 up to Day 12 of Period 2; Part 2: Day 1 of Period 1 up to Day 8 of Period 2
Population: All participants who received at least one dose of the study drug(s) were included in the safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Soticlestat 300 mg Alone | Part 1: Itraconazole 200 mg Alone | Part 1: Soticlestat 300 mg + Itraconazole 200 mg | Part 2: Soticlestat 300 mg Alone | Part 2: Mefenamic Acid 500 mg and 250 mg | Part 2: Soticlestat 300 mg + Mefenamic Acid 500 mg and 250 mg
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14
Participants | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Parts 1 and 2: Number of Participants With Clinically Significant Abnormal Values for Electrocardiogram (ECG)
Time Frame: Part 1: Day 1 of Period 1 up to Day 12 of Period 2; Part 2: Day 1 of Period 1 up to Day 8 of Period 2
Population: All participants who received at least one dose of the study drug(s) were included in the safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Soticlestat 300 mg Alone | Part 1: Itraconazole 200 mg Alone | Part 1: Soticlestat 300 mg + Itraconazole 200 mg | Part 2: Soticlestat 300 mg Alone | Part 2: Mefenamic Acid 500 mg and 250 mg | Part 2: Soticlestat 300 mg + Mefenamic Acid 500 mg and 250 mg
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14
Participants | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Parts 1 and 2: Number of Participants With Suicidal Ideation or Suicidal Behavior as Measured Using Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS is an interview-based rating scale to systematically assess any suicidality, suicidal behavior, or suicidal ideation. Any suicidality is emergence of any suicidal ideation or suicidal behavior. Any suicidal behavior was indicated when response was "yes" for any these questions- actual attempted to suicide, engaged in non-suicidal self-injurious behavior, interrupted attempt, aborted attempt, preparatory acts. Any suicidal ideation was indicated when response was "yes" for any of these questions- wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with methods without intent to act or some intended to act, without specific plan or with specific plan and intended to suicide.
Time Frame: Part 1: Day 1 of Period 1 up to Day 12 of Period 2; Part 2: Day 1 of Period 1 up to Day 8 of Period 2
Population: All participants who received at least one dose of the study drug(s) were included in the safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Soticlestat 300 mg Alone | Part 1: Itraconazole 200 mg Alone | Part 1: Soticlestat 300 mg + Itraconazole 200 mg | Part 2: Soticlestat 300 mg Alone | Part 2: Mefenamic Acid 500 mg and 250 mg | Part 2: Soticlestat 300 mg + Mefenamic Acid 500 mg and 250 mg
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14
Participants | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: TEAEs were adverse events (AE) that started from Day 1 of Period 1 up to 15 days after the last dose of soticlestat in Period 2 (up to Day 20 of Period 2) in Part 1; and from Day 1 of Period 1 up to 15 days after the last dose of soticlestat in Period 2 (up to Day 17 of Period 2) in Part 2
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Part 1: Soticlestat 300 mg Alone | Part 1: Itraconazole 200 mg Alone | Part 1: Soticlestat 300 mg + Itraconazole 200 mg | Part 2: Soticlestat 300 mg Alone | Part 2: Mefenamic Acid 500 mg and 250 mg | Part 2: Soticlestat 300 mg + Mefenamic Acid 500 mg and 250 mg
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 1/14 | 2/14 | 3/14 | 1/14 | 0/14 | 3/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Soticlestat 300 mg Alone (N=14) | Part 1: Itraconazole 200 mg Alone (N=14) | Part 1: Soticlestat 300 mg + Itraconazole 200 mg (N=14) | Part 2: Soticlestat 300 mg Alone (N=14) | Part 2: Mefenamic Acid 500 mg and 250 mg (N=14) | Part 2: Soticlestat 300 mg + Mefenamic Acid 500 mg and 250 mg (N=14)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2021-08-23): https://cdn.clinicaltrials.gov/large-docs/49/NCT05064449/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT05064449/SAP_001.pdf